CLINICAL TRIAL: NCT06994559
Title: Investigating the Synergistic Potential of Music as an Adjunct to Ketamine Therapy for Chronic Noncancer Pain
Brief Title: Music as an Adjunct to Ketamine Therapy for Chronic Pain
Acronym: MusKiP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Mathieu Roy, Associate Professor, McGill University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Music-Ketamine
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain; Chronic Noncancer Pain
Keywords: Chronic pain; Ketamine; Music
MeSH Terms: conditions — Chronic Pain | interventions — SIR1 protein, S cerevisiae

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Preferred-Therapist-Silence (Other): Participants in this arm will be exposed to 1) Preferred music, 2) Therapist-selected music and 3) Silence in this order
  Interventions: Other: Preferred Music; Other: Therapist-selected Music; Other: Silence
- Preferred-Silence-Therapist (Other): Participants in this arm will be exposed to 1) Preferred music, 2) Silence, and 3) Therapist-selected music, in this order
  Interventions: Other: Preferred Music; Other: Therapist-selected Music; Other: Silence
- Therapist-Preferred-Silence (Other): Participants in this arm will be exposed to 1) Therapist-selected music, 2) Preferred music, 3) Silence, in this order
  Interventions: Other: Preferred Music; Other: Therapist-selected Music; Other: Silence
- Therapist-Silence-Preferred (Other): Participants in this arm will be exposed to 1) Therapist-selected music, 2) Silence, and 3) Preferred music, in this order
  Interventions: Other: Preferred Music; Other: Therapist-selected Music; Other: Silence
- Silence-Therapist-Preferred (Other): Participants in this arm will be exposed to 1) Silence, 2) Therapist-selected music, and 3) Preferred music, in this order
  Interventions: Other: Preferred Music; Other: Therapist-selected Music; Other: Silence
- Silence-Preferred-Therapist (Other): Participants in this arm will be exposed to 1) Silence, 2) Preferred music, and 3) Therapist-selected music, in this order
  Interventions: Other: Preferred Music; Other: Therapist-selected Music; Other: Silence

INTERVENTIONS:
Other: Preferred Music — The self-selected preferred music intervention will expose participants to music chosen based on personal tastes. Patients will be instructed to compile a playlist lasting approximately 1 hour, but preferably over 1 hour (to avoid repetition or moments without music) of their favorite music. They will be instructed to select songs that they find extremely pleasurable to listen to. Participants will be instructed to select songs that will have a higher likelihood to facilitate relaxation and introspection. This does not need to be an all-time favorite selection, but rather the music that they currently enjoy listening to the most.
Other: Therapist-selected Music — The therapist-selected music intervention will expose participants to a curated playlist specifically designed for psychedelic treatment by expert Music Therapists, which was used in a previous study to investigate the additive hemodynamic effects of music during ketamine infusions for depression. Patients will be randomly exposed to one of 9 available playlists, all containing songs without lyrics.
Other: Silence — The silence intervention will expose patients to the same therapeutic procedures, in the same room and context, and with the same noise-cancelling headphones. The purpose is to cancel any potentially perturbing background noise, as no music will be played.

SUMMARY:
Intravenous (IV) ketamine is a treatment option for patients with chronic pain that does not respond to standard therapies, primarily working by blocking NMDA receptors in the brain. Beyond pain relief, ketamine can produce dissociative sensations, classifying it as an atypical psychedelic or mind-altering drug, and may enable patients to reprocess their pain similarly to experiences with traditional psychedelics. At the Montreal General Hospital's pain clinic, the investigators have observed patients frequently listening to music during ketamine infusions, and recent research indicates that music-especially when self-selected by patients-might provide additional pain-relieving benefits by influencing central mechanisms related to pain perception and interpretation. This intersection of music and pain relief is garnering substantial scientific interest as recent advances provide more insight into the neuroscience of music and its effects on brain regions involved in emotion, sensation, memory, and pain.

This study aims to investigate the effects of music on chronic pain patients undergoing IV ketamine infusions at the Alan Edwards Pain Management Unit (AEPMU), specifically to determine whether the choice of music affects the intensity and duration of ketamine-induced pain relief. During the infusion (lasting 1 hour), patients will listen to a playlist delivered through specialized headphones, which will either consist of their own selected music (preferred music), music chosen by a music therapist, or no music at all, in a randomized order. Patients will track their pain levels throughout the infusion period and in the intervals between treatments (5 weeks) using standardized pain assessment tools. Additionally, the investigators will assess the subjective experiences of ketamine through interviews and qualitative analysis, while documenting and summarizing any adverse effects.

The investigators hypothesize that listening to preferred music will enhance both the intensity and duration of pain relief from IV ketamine. To test this, the investigators will recruit patients already receiving repeated IV ketamine infusions for pain management at the AEPMU clinic. The first infusion will take place under usual conditions to establish a baseline. The infusions will occur in a dedicated room equipped with audio technology to ensure an immersive music experience.

DETAILED DESCRIPTION:
Chronic pain impacts nearly eight million Canadians, with many suffering from moderate to severe pain for over a decade. Traditional treatments often fail, prompting researchers to explore alternatives like intravenous (IV) ketamine infusions, initially developed as an anesthetic and now considered for conditions such as Complex Regional Pain Syndrome (CRPS) and fibromyalgia. Short-term benefits of ketamine for pain relief have been observed, but its long-term effects, optimal dosages, and safety profiles remain under investigation. Ketamine's psychedelic properties have shown potential in treating psychiatric conditions, suggesting it might alter patient's psychological outlook on their pain.

This study aims to investigate the potential synergistic effects of IV ketamine infusions combined with self-selected music on chronic noncancer pain. A total of 25 patients from the Alan Edwards Pain Management Unit (AEPMU) will participate in a pragmatic randomized crossover controlled trial involving four ketamine infusion sessions, each lasting one hour with a dosage of 0.5 mg/kg. The sessions will include a baseline control session with treatment as usual, and three different conditions: self-selected music, therapist-selected music, and silence. All participants will undergo the same therapeutic procedures in a controlled environment, with noise-cancelling headphones and dim lighting, to standardize the experience.

Participants will create personal music playlists lasting at least an hour, comprising songs that they find highly pleasurable and conducive to relaxation. Alternatively, they will be exposed to therapist-selected playlists designed specifically for psychedelic therapy or silence, ensuring a controlled setting with no background noise. The study will also require participants to engage with their music playlist or silence for one day each week, in a relaxed setting, to revisit their infusion experience.

To assess the effects, both quantitative and qualitative data will be collected, including pain intensity, mood, sleep, cognitive flexibility, and symptoms of anxiety and depression. Participants will undergo semi-structured interviews one week post-infusion to evaluate patient benefits and any adverse effects of the ketamine and music interventions. This innovative approach seeks to enhance the understanding of how music can optimize the therapeutic potential of ketamine infusions, offering a novel avenue for managing chronic pain where conventional treatments have proven inadequate.

The investigators anticipate that these findings will help optimize the use of IV ketamine at the AEPMU and in other settings where this treatment is available.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic (3 months) pain of noncancerous origin, including chronic primary and secondary pain conditions, irrespective of its mechanistic contributors (nociceptive, neuropathic, or nociplastic), and of moderate to severe intensity (rated ≥ 4 in a 0-10 scale);
* Participants must have been prescribed IV ketamine treatment at the AEPMU, based on their treating clinician's assessment and judgment;
* Prior their participation in the study, all Participants must have undergone at least one ketamine IV session in the AEPMU clinical setting, which was well tolerated and did not reveal any important adverse effects, and which is expected to be repeated;
* Be able to use an electronic device (e.g., computer, tablet, smartphone) to complete questionnaires and diaries. For patients who may not possess such a device, a smartphone will be loaned for the duration of the study;
* No contraindication for intravenous ketamine treatment, including: poorly controlled cardiovascular disease, pregnancy or current or past history of psychosis, moderate to severe hepatic disease, elevated intracranial or extraocular pressure, and current or past history of substance abuse;
* Abstention from consuming grapefruit juice on the day of the ketamine infusions as it may alter the metabolism of ketamine;

Exclusion Criteria:

* Low tolerability or ineffectiveness of previous intravenous treatment or ketamine infusions;
* Current diagnosis or treatment for cancer;
* Significant hearing impairment not improved with hearing aids and/or sound amplification or unwillingness to listen to music during treatment;
* Known intellectual disability or autism spectrum disorder;
* Known risk factors for intracranial hemorrhage, including previous significant trauma, known aneurysm, or previous neurosurgery;
* Evidence of clinically relevant disease, e.g., renal or hepatic impairment, significant coronary artery disease (myocardial infarct within a year prior to initial randomization), cerebrovascular disease, viral hepatitis B or C, acquired immunodeficiency syndrome or history of seizure disorder;
* Prior or current (i.e., past-year) history of substance use disorder (except for caffeine or nicotine use disorder) as defined by DSM-5 criteria;
* Acute psychotic or suicidal ideation symptoms, as judged by the referring clinician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | From baseline to 24 hours after each ketamine session
  Pain intensity assessed using a 0-10 visual rating scale anchored at 0 (absence of pain) and 10 (maximum pain imaginable). Participants will rate their average pain intensity in the previous 24 hours.

SECONDARY OUTCOMES:
In-session Pain intensity | Immediately before and after each ketamine session
  Pain intensity assessed using a 0-10 visual rating scale anchored at 0 (absence of pain) and 10 (maximum pain imaginable). Participants will rate their current pain intensity.
In-session Pain unpleasantness | Immediately before and after each ketamine session
  Pain unpleasantness assessed using a 0-10 visual rating scale anchored at 0 (absence of pain) and 10 (most unpleasant pain imaginable). Participants will rate their current pain intensity.
Duration of pain relief | From baseline to the end of each condition (5 weeks) daily for one week, then weekly
  Duration of pain relief will be assessed based on repeated self-reported pain intensity ratings using a 0-10 visual rating scale, collected at multiple time points over a 5-week follow-up period. This outcome will capture how long participants experience sustained reductions in pain following each intervention condition.
Brief Pain Inventory (pain interference) | From baseline to the end of each condition (5 weeks)
  Pain interference will be assessed using an 7-item questionnaire (Brief Pain Inventory, score range 0 to 10 per item, 0 to 70 in total).
Brief Pain Inventory (number of pain sites) | From baseline to the end of each condition (5 weeks)
  The number of body sites in which participants report pain will be assessed using a body map with up to 30 potential body sites (Brief Pain Inventory).
Pain Catastrophizing Scale (PCS) | From baseline to the end of each condition (5 weeks)
  Pain catastrophizing thoughts and beliefs will be assessed using a 13-item questionnaire (PCS, score range 0 to 52)
Hospital Anxiety and Depression Scale (HADS) | From baseline to the end of each condition (5 weeks)
  Anxiety and depression symptoms will be assessed using a 14-item questionnaire (HADS, score range 0 to 42), with separate subscales for anxiety (HADS-A) and depression (HADS-D), each ranging from 0 to 21.
Positive and Negative Affect Scale (PANAS) | From baseline to the end of each condition (5 weeks)
  Positive and negative affect will be assessed using a 20-item questionnaire (PANAS, score range 20 to 100), with separate subscales for positive affect (PA) and negative affect (NA), each ranging from 10 to 50.
Multidimensional Psychological Flexibility Inventory (MPFI), short form | From baseline to the end of each condition (5 weeks)
  Cognitive and behavioral flexibility will be assessed using a 24-item questionnaire (MPFI-24, score range 24 to 120), with separate subscales for cognitive and behavioral flexibility, each ranging from 12 to 60.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Ware, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Mathieu Roy, PhD, Principal Investigator — McGill University
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
IPD will be share upon reasonable request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be share upon reasonable request
Access Criteria: IPD will be share upon reasonable request

REFERENCES:
- [Background] Sorensen J, Bengtsson A, Backman E, Henriksson KG, Bengtsson M. Pain analysis in patients with fibromyalgia. Effects of intravenous morphine, lidocaine, and ketamine. Scand J Rheumatol. 1995;24(6):360-5. doi: 10.3109/03009749509095181. PMID 8610220
- [Background] Olofsen E, Kamp J, Henthorn TK, van Velzen M, Niesters M, Sarton E, Dahan A. Ketamine Psychedelic and Antinociceptive Effects Are Connected. Anesthesiology. 2022 May 1;136(5):792-801. doi: 10.1097/ALN.0000000000004176. PMID 35188952
- [Background] Lunde SJ, Vuust P, Garza-Villarreal EA, Vase L. Music-induced analgesia: how does music relieve pain? Pain. 2019 May;160(5):989-993. doi: 10.1097/j.pain.0000000000001452. No abstract available. PMID 30507782
- [Background] Greenway KT, Garel N, Goyette N, Turecki G, Richard-Devantoy S. Adjunctive music improves the tolerability of intravenous ketamine for bipolar depression. Int Clin Psychopharmacol. 2021 Jul 1;36(4):218-220. doi: 10.1097/YIC.0000000000000363. PMID 33902087
- [Background] Greenway KT, Garel N, Dinh-Williams LL, Beaulieu S, Turecki G, Rej S, Richard-Devantoy S. Music as an Intervention to Improve the Hemodynamic Response of Ketamine in Depression: A Randomized Clinical Trial. JAMA Netw Open. 2024 Feb 5;7(2):e2354719. doi: 10.1001/jamanetworkopen.2023.54719. PMID 38315489
- [Background] Garza-Villarreal EA, Pando V, Vuust P, Parsons C. Music-Induced Analgesia in Chronic Pain Conditions: A Systematic Review and Meta-Analysis. Pain Physician. 2017 Nov;20(7):597-610. PMID 29149141

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-05-20): https://cdn.clinicaltrials.gov/large-docs/59/NCT06994559/SAP_000.pdf